CLINICAL TRIAL: NCT01802086
Title: Emla-Cream as Pain Relief During Pneumococcal Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beatrice Olsson Duse (Other)
Responsible Party: Sponsor-Investigator, Beatrice Olsson Duse, RN, Sormland County Council, Sweden
Organization: Sormland County Council, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SormlandCC; 2010-021406-38 (EudraCT Number)
Record Dates: First submitted 2012-10-31; First posted 2013-03-01 (Estimated); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Children; Pain
Keywords: Children; Pain; Vaccination; Emla; Pneumococcal; Pain scale
MeSH Terms: conditions — Pain | interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine; Prilocaine; Glycerol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Emla-cream (Active Comparator): Dose: 1 g Emla-cream, 1 hour.
  Interventions: Drug: Emla-cream
- Miniderm cream (Placebo Comparator): Dose: 1 g Miniderm-cream, 1 hour.
  Interventions: Drug: Miniderm cream

INTERVENTIONS:
Drug: Emla-cream — Topical anaesthetic
  Other Names: Studied drug: Emla-Cream, lidocaine and prilocaine
  Arms: Emla-cream
Drug: Miniderm cream — Topical
  Other Names: Placebo: Miniderm cream containing 20 % glycerol, non-pharmacological agent
  Arms: Miniderm cream

SUMMARY:
The aim of this intervention study is to compare the efficacy of Emla cream as a pain relief or no pain relief in connection to the first pneumococcal vaccination at the age of three months in Child health care.

Primary objective

1.Leads Emla cream as pain relief to children in connection with pneumococcal vaccination at the age of three months to lower pain scores in the use of five items; Face, Legs, Activity, Cry, Consolability (FLACC scale) as a pain measurement instrument?

DETAILED DESCRIPTION:
The aim of this intervention study is to compare the efficacy of Emla cream as a pain relief or no pain relief in connection to the first pneumococcal vaccination at the age of three months in Child health care.

Primary objective

1. Leads Emla cream as pain relief to children in connection with pneumococcal vaccination at the age of three months to lower pain scores in the use of FLACC scale as a pain measurement instrument?

   Secondary objectives
2. Leads Emla cream as pain relief in connection with pneumococcal vaccination to any difference in the child's heart rate response and saturation?
3. Leads Emla cream as pain relief that it takes longer before the baby starts crying and does the child cry for a shorter time in connection with vaccination?

Method: The study is randomised and singleblind. The study involves 72 children who are 3 months old. 36 children will receive Emla-cream and 36 children will receive placebo-cream.

This study will lead to new knowledge about Emla cream and pneumococcal vaccination. The study will give new knowledge how painful pneumococcal vaccination is for the children. If the study shows that Emla cream don´t give enough pain relief during pneumococcal vaccination more studies should be done with other pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, born vaginally or by cesarean section after 37 weeks of gestation, who were not admitted to the neonatal unit. Children should only have been with the newborn screening performed routinely at the hospital.

Exclusion Criteria:

* Baby delivered by vacuum extraction or forceps. Children born before gestational week 37. Children in neonatal care and subjected to other testing than newborn screening. Shoulder dystocia. Children susceptible to methaemoglobinaemia in glucose 6-phosphate dehydrogenase deficiency, congenital or idiopathic methemoglobinemia. Children with atopic dermatitis.

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bartocci, MD, PhD, Principal Investigator — Astrid Lindren Children´s Hospital
Locations (1):
- Healthcare center Mariefred/Strängnäs, Mariefred, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Emla-cream: Dose: 1 g Emla-cream, 1 hour.
  Emla-cream: Topical anaesthetic
  36 infants received Emla (intervention)
- Miniderm Cream: Dose: 1 g Miniderm cream, 1 hour.
  Miniderm cream: Topical
  34 infants received Miniderm Cream (placebo).
Period: Overall Study
Arm/Group | Emla-cream | Miniderm Cream
Started | 36 | 36
Completed | 36 | 36 (After statistics we excluded from the analysis two subjects.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emla-cream | Miniderm Cream | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 36 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 13 | 19 | 32

OUTCOME MEASURES:

1. Primary Outcome: Measuring the Effect of Emla Cream on Pain Perception During Pneumococcal Vaccination Measured With Five Items; Face, Legs, Activity, Cry, Consolability (FLACC Scale).
Description: The effect of Emla cream on pain perception during pneumococcal vaccination was measured by FLACC scale that includes five items; Face, Legs, Activity, Cry, Consolability. FLACC scale i a qualitative behavioural scale used for pain assesment and has been validated for use in infants aged 2 months to 7 years. Each item (Face, Legs, Activity, Cry and Consolability) can give 0,1 or 2 points according to the description included in the FLACC scale. The total summarised pain score can range between 0-10 points. A higher pain-score indicate more pain, which means a worse outcome.
  FLACC scale was measured before and after vaccination and compared between the groups (Emla-cream vs Miniderm cream).
Time Frame: Before vaccination and after vaccination, up to three minutes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Emla-cream | Miniderm Cream
Number analyzed (Participants) | 36 | 36
score on a scale
  FLACC score before vaccination | 0 [0 to 2] | 0 [0 to 4.5]
  FLACC score after vaccination | 7 [6 to 9] | 9 [7 to 9]

2. Secondary Outcome: Pain Perception Measured With Latency Time to Cry and Total Crying Time.
Description: Latency time to cry (scored in seconds):
  * how long does it takes until the baby starts to cry after vaccination was performed (the longer it takes until the baby starts to cry indicate less pain, a better outcome). Min- or maximum values is not applicable.
  Total crying time (scored in seconds):
  * how long time is the baby crying after vaccination was performed (the longer time the baby is crying indicate more pain, a worse outcome). Min- or maximum values is not applicable.
Time Frame: Before vaccination and after vaccination, up to three minutes.
Population: We analysed for how long time it takes until the baby starts to cry and for how long time the baby is crying.
Measure: Mean (Standard Deviation); unit: Time in seconds
Arm/Group | Emla-cream | Miniderm Cream
Number analyzed (Participants) | 36 | 36
Time in seconds
  Latency time to cry (seconds) | 2.77 (0.80) | 2.05 (0.978)
  Total crying time (seconds) | 78.74 (45.866) | 100.44 (73.307)

3. Secondary Outcome: Heart Rate (Beats Per Minute) Before and After Vaccination
Description: Heart rate before and after vaccination (beats per minute), higher values indicate more pain, a worse outcome. Min and max values are not applicable.
Time Frame: Before vaccination and after vaccination, up to three minutes
Population: We analysed the babies heart rate (beats per minute) before and after vaccination.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Emla-cream | Miniderm Cream
Number analyzed (Participants) | 36 | 36
beats per minute
  Beats per minute before vaccination | 148.31 (17.33) | 147.93 (17.95)
  Beats per minute after vaccination | 159.59 (15.53) | 160.46 (17.36)

4. Secondary Outcome: Saturation Before and After Vaccination.
Description: Oxygen saturation before and after vaccination (0-100%), a lower value indicate more pain, a worse outcome
Time Frame: Before vaccination and after vaccination, up to three minutes
Population: We analysed the babies oxygen saturation before and after vaccination.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Emla-cream | Miniderm Cream
Number analyzed (Participants) | 36 | 36
percentage of oxygen saturation
  Before vaccination | 99.59 (0.82) | 99.78 (0.43)
  After vaccination | 98.86 (1.22) | 98.76 (2.06)

ADVERSE EVENTS:
Time Frame: The follow-up time was one week. During the data collection, no adverse events occurred.
Description: No definitions differed to ClinicalTrials.gov.
Arm/Group | Emla-cream | Miniderm Cream
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No